CLINICAL TRIAL: NCT06970535
Title: Breastmilk Composition and Microbial Profile in the Growth and Development of Healthy Term-born Infants
Status: Withdrawn | Type: Observational
Why Stopped: Pandemic related complications made the study no longer feasible.
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Unity Health (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000067542
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breastmilk Collection; Childhood Obesity; Childhood Asthma; Allergy
Keywords: maternal metabolic status; term-born infants; breastmilk composition
MeSH Terms: conditions — Breast Milk Expression; Pediatric Obesity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human breastmilk samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An increasing number of children are developing non-communicable diseases that carry immediate and long-term significant societal and economic impacts. Thus, its prevention is imperative with early interventions, such as those that may fall within the first 1000 days, likely to yield better outcomes. The first 1000 days of life represent a period of rapid development sensitive to influences that may be leveraged to promote healthy growth. Breastfeeding is one such modifiable factor. Observational studies have shown that breastfeeding may be associated with reductions in chronic conditions, though its mechanism remains unknown. The complexity of these relationships is furthered by studies showing maternal metabolic status may alter breastmilk composition. Accordingly, this study aims to evaluate the influence of maternal metabolic status on breastmilk composition and assess associations between breastmilk composition and common noncommunicable diseases in childhood.

DETAILED DESCRIPTION:
This project will be completed within TARGet Kids! (The Applied Research Group for Kids), a paediatric primary care research network (NCT01869530). Mother-infant dyads will be recruited and a breastmilk sample obtained at three months of age. Children will then be seen as part of routine care for the next five years to track growth, health and development. This study will provide the opportunity of prospectively following term-born Canadian children to understand the relationship between breastfeeding patterns and child health, its potential underlying mechanisms and how breastmilk composition is modified by maternal metabolic status, which altogether can be used to help set children on optimal developmental trajectories.

STUDY OBJECTIVES:

1. To evaluate the influence of maternal metabolic status, on breastmilk composition (energy, macronutrient and micronutrient content and microbial profile) at three months post-partum.

   * Maternal metabolic status will be characterized by: maternal obesity (measured), diabetes, hypertension and gestational weight gain (self-reported).
2. To assess the associations between breastmilk composition and obesity, asthma and allergy in the children longitudinally to five years of age.

ELIGIBILITY:
Inclusion Criteria:

* The child is a participant in the TARGet Kids! (The Applied Research Group for Kids) study (NCT01869530)
* The child is between two and four months of age at recruitment.
* The child is healthy.
* Child is fed exclusively mother's milk and has not received any infant formula, cow's milk, juice, tea, or solids in the two weeks prior to recruitment.
* The mother of the child is present at the time of recruitment.

Exclusion Criteria:

* The child was born at <37 weeks gestation.
* The child has been diagnosed with a health condition affecting growth (e.g. failure to thrive, cystic fibrosis).
* The child has been diagnosed with any acute or chronic conditions.
* The family of the child is unable to communicate in English.

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mother-infant dyads will be recruited prospectively within the TARGet Kids! cohort. According to current TARGet Kids! study procedures (NCT01869530), initial contact with families is made by email or letter, from the child's paediatric clinic, two weeks prior to the scheduled visit. Families will also be made aware of the study through posters and informal conversations during early postnatal well-child visits.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2026-01-11 (Estimated); Study Completion 2026-01-11 (Estimated)

PRIMARY OUTCOMES:
Breastmilk composition - Total Energy | 3-months postpartum
  Total energy content of breastmilk samples measured using a mid-infrared human milk analyzer
Breastmilk composition - Macronutrients | 3-months postpartum
  Macronutrient content of breastmilk samples (fat, protein & carbohydrate) measured using a mid-infrared human milk analyzer
Breastmilk composition - Micronutrients | 3-months postpartum
  Micronutrient content of breastmilk samples (examples include vitamin B12 and choline)
Breastmilk composition - Microbial profile | 3-months postpartum
  Microbial profile of breastmilk samples using 16S rRNA gene sequencing and PCR amplification

SECONDARY OUTCOMES:
Child growth | 3-months postpartum to 5-years of age
  Weight and length/height measured at well-child visits to calculate BMI age- and sex-specific z-scores, annually until 5-years of age
Childhood allergies | 3-months postpartum to 5-years of age
  Measured by parental-report via questionnaire at well-child visits annually until 5-years of age
Childhood asthma | 3-months postpartum to 5-years of age
  Measured by parental report via questionnaire at well-child visits annually until 5-years of age

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD, RD, Principal Investigator — The Hospital for Sick Children; Catherine Birken, MD,MSc,FRCPC, Principal Investigator — The Hospital for Sick Children; Jonathon Maguire, MD,MSc,FRCPC, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - Unity Health Toronto, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No